CLINICAL TRIAL: NCT01792115
Title: Treatment for Non-Alcoholic Fatty Liver With Different Doses of Vitamin E
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 130002; 13-DK-0002 (Other: NIH Clinical Center)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-03-05

CONDITIONS: Fatty Liver
Keywords: Fatty Liver; Alpha-Tocopherol; Vitamin E; Non-Alcoholic Steatohepatitis
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Vitamin E; Diet; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vit E 200 IU/d (Active Comparator): Subjects randomized to vitamin E 200 IU/day for 24 weeks; invited to optional extension of open- label vitamin E 800 IU /day for up to 120 weeks following the initial 24 week period.
  Interventions: Drug: Vitamin E 200 IU/d; Behavioral: Diet and Exercise
- Vitamin E 400 (Active Comparator): Subjects randomized to vitamin E 400 IU/day for 24 weeks; invited to optional extension of open- label vitamin E 800 IU/day for up to 120 weeks following the initial 24 week period.
  Interventions: Drug: Vitamin E 400 IU/d; Behavioral: Diet and Exercise
- Vitamin E 800 (Active Comparator): Subjects randomized to vitamin E 800 IU /day for 24 weeks; invited to optional extension of open- label vitamin E 800 IU /day for up to 120 weeks following the initial 24 week period.
  Interventions: Drug: Vitamin E 800 IU/d; Behavioral: Diet and Exercise

INTERVENTIONS:
Drug: Vitamin E 200 IU/d — Supplement-low dose
  Arms: Vit E 200 IU/d
Drug: Vitamin E 400 IU/d — Supplement-intermediate dose
  Arms: Vitamin E 400
Drug: Vitamin E 800 IU/d — Supplement High Dose
  Arms: Vitamin E 800
Behavioral: Diet and Exercise — Diet and Exercise for all Arms of the study at baseline

SUMMARY:
Background:

* Non-alcoholic fatty liver disease (NAFLD) is an excess accumulation of fat in the liver cells. It is associated with obesity, high blood pressure, high cholesterol, and diabetes. Some people with NAFLD only have excess fat in the liver. However, other people may develop a worse form of NAFLD with liver injury and scarring. This form, called non-alcoholic steatohepatitis (NASH), can lead to liver failure, liver cancer, and death. Not much is known about why some people develop NASH and others do not.
* Lifestyle changes such as diet, exercise, and weight loss can decrease the liver damage in NAFLD. Some studies show that vitamin E can also help treat NAFLD. The dose of vitamin E used in these studies is almost 40 times the recommended amount of vitamin E intake from food. It is unclear whether a lower dose could achieve the same effect. Researchers also want to study how vitamin E works at different doses to treat NAFLD.

Objectives:

* To find out the most effective dose of vitamin E to treat NAFLD.
* To gain a better understanding of how NAFLD and NASH develop, and predict who will respond to treatment.

Eligibility:

- Individuals at least 18 years of age with suggestion of non-alcoholic fatty liver disease.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* For the first 12 weeks of the study, participants will meet with a nutritionist. They will have personalized diet and exercise plans. Treatment will be monitored with diaries and questionnaires to fill out at home. Participants will also wear a pedometer to measure physical activity.
* After the 12-week period, participants will have a full physical examination with the following tests:
* Blood tests
* Glucose tolerance tests
* Imaging studies (DEXA scan and magnetic resonance imaging)
* Liver and fatty tissue biopsy
* Two weeks after the tests, participants will start vitamin E treatment. They will take up to two pills a day, taken with fat-containing foods.
* 4 weeks after starting treatment they will have a repeat full evaluation with imaging tests, blood work, and liver and fat biopsies.
* Participants who are taking vitamin E will take it for up to 120 weeks. They will have monitoring visits every 8 to 12 weeks. At the end of 120 weeks, they will have another full evaluation, with imaging tests, blood work, and liver and fat biopsies.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common cause for liver test abnormalities in the western world, and an increasingly rising cause for liver-related morbidity and mortality. Vitamin E, a fat-soluble anti-oxidant was recently found to be an effective treatment for NAFLD; however, its mechanism of action is unclear. In a controlled clinical trial vitamin E treatment was shown to significantly reduce the hepatic fat burden, suggesting mechanisms other than reducing oxidative stress are involved. Furthermore, the optimal dose of vitamin E to treat NAFLD is unknown.

We propose a phase IIa study to determine the optimal dose of vitamin E and its mechanism and site of action. In this study we aim to enroll up to 90 patients with NAFLD. Initially, all patients will undergo 12 weeks of intensive lifestyle modification. Following that, all patients will be randomized to treatment with 3 different doses of natural vitamin E (rrr- -tocopherol at 200, 400 or 800 IU/d) for 24 weeks. The primary end points for efficacy are normalization of liver enzymes and reduction in liver fat contents by magnetic resonance spectroscopy. Patients will undergo liver and adipose tissue biopsies before vitamin E treatment and after 4 weeks of therapy, and the biopsy samples will be used to measure changes in gene expression and markers of oxidative stress. This will be coupled with extensive phenotyping before and after treatment using serological, radiological and dynamic endocrine testing and is aimed at finding the dose-response characteristics of vitamin E in NAFLD, and allowing us to understand the mechanism of its action.

After 24 weeks of randomized treatment, all patients will be switched to a dose of 800 IU/ml and will continue treatment for up to 30 months, at the end of which another liver biopsy will be performed. From this phase we will assess the effects of dose increase of vitamin E on liver enzymes and fat content, and will determine the effect of long-term treatment on histological outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:

Clinical suspicion of NAFLD, defined by the presence of at least two of the following criteria:

* Suggestion of liver fat by an imaging study (ultrasound, CT scan, MRI or MR spectroscopy) performed in the 6 months prior to enrollment.
* Elevated aminotransferase levels (ALT > 31 U/L for men or > 19 U/L for women, or AST > 30 U/L) on at least two occasions in the 6 months preceding enrollment.
* Presence of the metabolic syndrome, defined according to the modified AHA/NCEP criteria as the presence of at least three of:

  * Abdominal obesity, defined as waist circumference > 102 cm for men or > 88 cm for women
  * Elevated triglycerides (> 150 mg/dL) or the use of medication to lower triglycerides
  * Reduced HDL cholesterol (< 40 mg/DL for men or < 50 mg/dL for women)
  * Elevated blood pressure (> 135/80 mmHg) or use of medication for hypertension
  * Elevated fasting glucose levels (> 100 mg/dL) or use of anti-diabetic medication

    * For the purpose of inclusion, the presence of overt diabetes mellitus type 2 will be considered equivalent to the presence of the metabolic syndrome, even if the other criteria are absent.
* Estimated average alcohol consumption < 30 g/d for men or < 20 g/d for women in the 6 months prior to enrollment and no binge-drinking behavior.
* Age > 18 years at enrollment
* Willingness to participate in the study

EXCLUSION CRITERIA:

* Chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV). Patients who were treated successfully for HCV and achieved sustained virological response can be eligible for enrollment > 18 months after treatment cessation. Patients who are inactive carriers of HBV (HBV DNA < 1000 copies/mL, HBeAg negative, Anti HDV negative) for at least 12 months prior to enrollment are also eligible. Patients receiving antiviral therapy are ineligible.
* Concomitant liver disease such as autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson s disease, alpha-1 antitrypsin deficiency.
* Presence of definite or probable drug-induced liver injury. In the case of lipid-lowering, anti-hypertensive or anti-diabetic medications that are suspected to cause elevation of aminotransferases, patients will be eligible if treatment is associated with stable enzyme levels for at least 6 months and inclusion criteria 1a. and 1c. are both present.
* Treatment with medications known to cause fatty liver disease such as atypical neuroleptics, tetracycline, methotrexate or tamoxifen
* Uncontrolled hypo- or hyperthyroidism.
* Decompensated advanced liver disease, defined as direct bilirubin > 0.5 g/dL, PT > 18, albumin < 3 g/dL, or history of ascites, encephalopathy, variceal bleeding, spontaneous bacterial peritonitis or liver transplant.
* Active coronary artery disease, defined as persistent angina pectoris, reversible ischemia on cardiac stress test or imaging, or the presence of significant coronary artery disease on imaging or catheterization. Patients with coronary artery disease that was treated by angioplasty or bypass surgery may be eligible if they have no evidence of active disease >= 1 year after intervention, can safely stop antiplatelet and anticoagulant medications before the performance of invasive procedures, and have adequate ventricular function as assessed by echocardiography or cardiology consultation. These patients will require cardiology consultation and clearance prior to enrollment.
* Congestive heart failure.
* Chronic kidney disease, with creatinine clearance < 60 ml/h.
* Uncontrolled diabetes mellitus. Patients may be enrolled if they have been on stable therapy with any anti-diabetic agent for at least 3 months prior to enrollment, are not foreseen by the physician treating their diabetes to require antidiabetic medication or dose changes during the trial and have an HbA1c <= 7.5% on enrollment.
* Treatment with vitamin E. Patients who are currently taking vitamin E as a supplement will be requested to stop for at least 3 months before becoming eligible for enrollment. Patients who are taking vitamin E for a medical indication other than NAFLD will not be eligible.
* Contraindication to or inability to undergo a liver biopsy.
* Patients who had a liver biopsy performed <= 2 years before enrollment, unless they are willing to undergo all of the trial biopsies, knowing that these biopsies are purely for research and are not clinically indicated. This will be clearly documented in the patients charts prior to enrollment.
* Patients with coagulopathy (PT/PTT values that are prolonged >= 3 seconds from the upper limit of the normal, including treatment with oral and parenteral anticoagulants), thrombocytopenia (<70,000), or platelet dysfunction will not be enrolled because of potential increase in risk of bleeding with vitamin E treatment. Antiplatelet agents taken for cardiovascular prevention will not exclude patients, unless they cannot be stopped safely for the performance of a liver biopsy.
* Maldigestion or malabsorption that can interfere with absorption of vitamin E including: steatorrhea of all causes, chronic pancreatitis, cystic fibrosis, short bowel syndrome, severe cholestasis, orlistat treatment and similar conditions
* Inability to swallow vitamin E capsules
* Allergy to vitamin E
* Alcohol or substance abuse within the past 12 months. Patients will be required to have an AUDIT score of 7 or less18, and drink no more than 14 drinks/week (for men) or 7 drinks/week (for women).
* For women of childbearing age, pregnancy or inability (or unwillingness) to practice contraception for the duration of the study or breast feeding.
* Inability to understand and give informed consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rotman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Podszun MC, Alawad AS, Lingala S, Morris N, Huang WCA, Rotman Y. Development of Subtle Iron Deficiency During Vitamin E Treatment For Metabolic Dysfunction-Associated Steatotic Liver Disease. J Diet Suppl. 2025;22(2):284-299. doi: 10.1080/19390211.2025.2465414. Epub 2025 Feb 17. PMID 39960325
- [Derived] Podszun MC, Alawad AS, Lingala S, Morris N, Huang WA, Yang S, Schoenfeld M, Rolt A, Ouwerkerk R, Valdez K, Umarova R, Ma Y, Fatima SZ, Lin DD, Mahajan LS, Samala N, Violet PC, Levine M, Shamburek R, Gharib AM, Kleiner DE, Garraffo HM, Cai H, Walter PJ, Rotman Y. Vitamin E treatment in NAFLD patients demonstrates that oxidative stress drives steatosis through upregulation of de-novo lipogenesis. Redox Biol. 2020 Oct;37:101710. doi: 10.1016/j.redox.2020.101710. Epub 2020 Sep 1. PMID 32920226
- [Derived] Podszun MC, Chung JY, Ylaya K, Kleiner DE, Hewitt SM, Rotman Y. 4-HNE Immunohistochemistry and Image Analysis for Detection of Lipid Peroxidation in Human Liver Samples Using Vitamin E Treatment in NAFLD as a Proof of Concept. J Histochem Cytochem. 2020 Sep;68(9):635-643. doi: 10.1369/0022155420946402. PMID 32867573
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-DK-0002.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Started | 7 | 7 | 8
Completed | 7 | 6 | 8
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800 | Total
Number analyzed (Participants) | 7 | 7 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (14.6) | 43.9 (9.3) | 48.4 (11.3) | 48.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 10
  Male | 2 | 4 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 5 | 14
  Not Hispanic or Latino | 2 | 3 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 3 | 2 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 5 | 14
Diabetes [Count of Participants; unit: Participants]
  Has Diabetes | 0 | 2 | 3 | 5
  No Diabetes | 7 | 5 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Biochemical: Number of Patients With Normal Transaminases at End of Treatment.
Description: Biochemical response defined as number of patients with normal transaminases AST <=32 or ALT <=35 U/L at end of treatment.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Number analyzed (Participants) | 7 | 6 | 8
Participants | 6 | 6 | 6

2. Primary Outcome: Physiological: Absolute Change in Liver Fat
Description: Physiological response defined as absolute change in liver fat measured by 1H-MRS
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percent liver fat
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Number analyzed (Participants) | 6 | 6 | 8
percent liver fat | -1.9 (9.6) | -7.6 (3.3) | -0.6 (5.2)

3. Secondary Outcome: Absolute Change in AST
Description: Absolute Change in AST [u/l] by week 24
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: u/l
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Number analyzed (Participants) | 7 | 6 | 8
u/l | -5.6 (11.1) | -1.8 (4.5) | -10.6 (16.7)

4. Secondary Outcome: Percent Change in AST
Description: Percent change in AST by week 24
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Number analyzed (Participants) | 7 | 6 | 8
percent | -0.15 (0.29) | -0.07 (0.21) | -0.24 (0.4)

5. Secondary Outcome: Absolute Change in ALT
Description: Absolute Change in ALT [u/l] by week 24
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: u/l
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Number analyzed (Participants) | 7 | 6 | 8
u/l | -8 (16.7) | -8.3 (10.7) | -22 (22)

6. Secondary Outcome: Percent Change in ALT
Description: Percent change in ALT by week 24
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Number analyzed (Participants) | 7 | 6 | 8
percent | -0.17 (0.44) | -0.19 (0.23) | -0.35 (0.27)

7. Secondary Outcome: Absolute Change in GGT
Description: Change in GGT by week 24 (U/L)
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: u/l
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Number analyzed (Participants) | 7 | 5 | 8
u/l | -6.1 (24.5) | -22.8 (50) | -11 (18.9)

8. Secondary Outcome: Percent Change in Liver Fat
Description: Percent change in liver fat by week 24
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percent of percent liver fat
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
Number analyzed (Participants) | 6 | 6 | 8
percent of percent liver fat | 0.33 (0.93) | -0.42 (0.18) | -0.10 (0.48)

ADVERSE EVENTS:
Time Frame: AE data were collected over 144 weeks, from starting treatment to completion of treatment.
Arm/Group | Vit E 200 IU/d | Vitamin E 400 | Vitamin E 800
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7 | 3/8
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vit E 200 IU/d (N=7) | Vitamin E 400 (N=7) | Vitamin E 800 (N=8)
Gastrointestinal Bleed (Gastrointestinal disorders) | 0 | 0 | 1
Diuretic-induced hypokalemia (Renal and urinary disorders) | 0 | 0 | 1
Diverticulitis with recto-vaginal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Hypertensive crisis (medication non-compliance) (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vit E 200 IU/d (N=7) | Vitamin E 400 (N=7) | Vitamin E 800 (N=8)
Depression (Psychiatric disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Headache/Migraine (Nervous system disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Viral gastroenteritis (Infections and infestations) | 1 | 0 | 0
Galactorrhea (Reproductive system and breast disorders) | 1 | 0 | 0
Breast cancer (Reproductive system and breast disorders) | 1 | 0 | 0
Hypertensive crisis (Cardiac disorders) | 1 | 0 | 0
Muscle tear (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Herpes Keratitis (Infections and infestations) | 0 | 1 | 0
Vasovagal (Cardiac disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Epistaxis (Vascular disorders) | 0 | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (post-anesthesia) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertriglyceridemia exacerbation (Vascular disorders) | 0 | 0 | 1
Jaw swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1
Iron deficiency or anemia (Blood and lymphatic system disorders) | 3 | 4 | 4
Overt gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT01792115/Prot_SAP_000.pdf